CLINICAL TRIAL: NCT03848377
Title: A Feasibility Study of a Novel Combined Automated EMG and SSEP Device (EPAD® 2.0) for Intraoperative Monitoring of Spinal Nerve Roots and Spinal Cord Function During Spine Surgery
Brief Title: EMG and SSEP Device (EPAD® 2.0) for Intraoperative Monitoring of Patient Undergoing Spinal Nerve Spine Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Jason Chui, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: 112933
Record Dates: First submitted 2019-02-19; First posted 2019-02-20 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Spine Disease; Neurological Disorder
Keywords: Spine surgery; Neuromonitoring; Evoked potential; electromyography; neurological injury
MeSH Terms: conditions — Spinal Diseases; Nervous System Diseases; Trauma, Nervous System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Automated EMG/SSEP monitored: In this study, all patients will be monitored for SSEP and EMG. For SSEP monitoring, surface adhesive electrodes will be used for both stimulation and recording. After an automatic impedance check, the baseline subcortical SSEP will be established at the beginning of each case, and the amplitude and latency of the waveforms will be measured. For EMG monitoring, 6 Surface electrodes will be attached to the same muscle groups of the conventional intraoperative neurophysiological monitoring machine. In each case, the Compound Muscle Action Potentials (CMAPs) of each muscle group will be monitored.
  As this is an observational study, no intervention is planned.

SUMMARY:
In patients undergoing spine surgery, spinal nerve roots and spinal cord are vulnerable to surgical insults especially for instrumentation and may lead to long term sequelae. The incidence of clinical peripheral neuropathy after cervical spine surgery has been reported up to 30%. Intraoperatively, spinal cord and nerves function can be monitored using electromyography (EMG) and somatosensory evoked potentials (SSEP) and thereby, intervention can be made to potentially reduce the incidence of adverse neurological sequelae. However, conventional EMG and SSEP monitoring requires presence of a trained EP technician, use of needle electrodes and currently bulky EP equipment and is thus not practical for routine clinical usage. In this study, the invesitgators will assess the clinical feasibility of using a novel miniaturized and automated EMG/SSEP device (EPAD® 2.0) in spine surgical patients.

DETAILED DESCRIPTION:
Purpose of Research: This study is a pilot study designed to assess the ability of a novel automated EMG/SSEP device (EPAD® 2.0) to detect intraoperative spinal nerve roots injury in patients undergoing spine procedures. The specific aims are:

1. to assess the clinical utility of using the EPAD® 2.0 automated device and its algorithm in monitoring spine surgery patients.
2. to identify any practical limitation of using EPAD® 2.0 automated device in spine surgery patients.

Hypothesis: the novel automated EPAD® 2.0 EMG/SSEP device is easy to use and apply in spine surgery patients

BACKGROUND Surgical injuries to the spinal nerve roots or spinal cords are not infrequent in spine surgery and the consequence can be devastating. Injured patients might present with radiculopathy, motor weakness, spinal cord compression, and postoperative neuropathic pain. In cervical spine surgery, cervical nerve roots injuries especially fifth cervical (C5) nerve root are not uncommon complications, potentially resulting in upper extremity paralysis. The incidence of C5 nerve root injury ranged to as high as 30%. The other spinal nerve roots (C6-8) can suffer from the same surgical injuries during the procedure but with much lower reported incidence than C5. Spinal nerve injuries typically occur during decompression for cervical myelopathy in both anterior and posterior approaches. In lumbosacral spine surgery, a recent review of the neurological injury found a pooled incidence of 5.7% (56 of 2783 patients; range: 0.46-24%), in which pedicle malposition accounted for one-fifth of the injuries.

A multimodality monitoring such as SSEP and EMG can be used in spine surgery to allow comprehensive monitoring of the spinal cord and nerve roots function and an attempt to reduce the risks of surgical injuries. Although the idea of closely monitoring of spinal cord and nerve roots function during high-risk cervical spine instrumentation procedure is appealing, the utilization of intraoperative neurophysiological monitoring is limited. One reason is the current requirements for a trained technician and for electrode placement and observation of monitoring SSSEP signals, the requirement for the use of needle electrodes for SSEP monitoring and specific training for a neurophysiologist in the interpretation of SSEP signals.

In attempt to resolve this problem, the investigators has been involved in developing an automated SSEP device (EPAD®, SafeOp Surgical, Hunt Valley, MD; FDA approved). The automated EPAD1.0 SSEP device the investigators are currently utilizing is miniaturized and incorporates a proprietary technology utilizing non-invasive electrode patches (rather than needle electrodes) and is based on an automated algorithm derived from real-time SSEP monitoring of over 100,000 surgical procedures. The investigators was the first to evaluate the clinical utility of this automated SSEP device in cardiac surgical and total shoulder arthroplasty patients. These pilot studies found that automated SSEP monitoring can be performed readily in a busy cardiac operating room, as well as in orthopedic surgery. The raw signal quality is reliable and comparable to the conventional SSEP machine. These results indicate that this device can eliminate the practical challenges of performing SSEP monitoring and confirmed its feasibility for routine use. The initial experience has enabled further development that has incorporated software updates based on off-line data-reiteration. This has also allowed progressive refinement of the automated analysis algorithm based on this recently acquired intraoperative SSEP data to progressively optimize the software for improved signal acquisition, enhanced artifact rejection and electrocautery suppression.

METHOD Study Design This will be a prospective cohort study aiming in assessing the ability of a novel automated EMG/SSEP device (EPAD® 2.0) to detect intraoperative spinal nerve root injury in patients undergoing spine procedures. All protocol procedures will be undertaken; however, as this is the first clinical trial of EPAD® 2.0, the initial series of up to 30 patients will be used for feasibility anticipating some possible minor software revisions and minor equipment modifications. Additionally, data obtained from this initial series of patients may be utilized to iteratively refine the data collection and analysis algorithms.

Standard Procedure After obtaining preoperative written consent, a brief neurological exam will be conducted. As is conventional, anesthesia will be induced using opioid/propofol and will be maintained with halogenated anesthetic agents and supplemented with an infusion of remifentanil at 0.01-0.2 mcg/kg/min or sufentanil at 0.15 to 0.5g/kg/hr. Muscle relaxants will only be given for intubation and no second dose will be given to enable EMG monitoring. After anesthesia induction with airway and vascular access secured, the patient will be positioned for the surgery. There is no change in routine (or standard) of care except the investigators will attach the EPAD 2.0 device to the patients. After the surgery, the patient will be extubated and transferred to PACU. In all patients, a complete neurological exam will be performed in PACU.

Study Procedure:

For SSEP monitoring, surface adhesive electrodes will be used for both stimulation and recording. Stimulating electrodes will be placed for stimulation of the dermatome that is at risk of injury (e.g. C5), median nerve or posterior tibal nerve. Recording surface electrodes will be placed on the cervical spine at the C2 level (C2), and the reference electrode was placed on the forehead. The pre-set stimulation frequency in the EPAD device is 4.7 Hz with a 300- microsecond pulse set at 50 to 70 mA and the signal averaging set at 300 cycles. After an automatic impedance check, the baseline subcortical SSEP will be established at the beginning of each case, and the amplitude and latency of the waveforms will be measured. The EPAD device automatically established the baselines.

For EMG monitoring, 6 Surface electrodes will be attached to the same muscle groups of the conventional intraoperative neurophysiological monitoring machine. The underlying skin will be prepared with 3M EKG skin abrasive tape (3M red dot 2236) to reduce the skin impedance. In each case, the Compound Muscle Action Potentials (CMAPs) of each muscle group will be monitored. The EMG monitoring can provide three main functions in spine surgery, which includes free-run EMG for detecting mechanical irritation to nerve root, triggered EMG for nerve root identification and pedicle screw placement assessment. All three EMG functions will be evaluated in this study.

Short Summary of Study Protocol:

1. Written informed consent
2. Focused neurological exam preoperatively
3. Placement of surface electrodes in OR
4. Monitoring during the spine procedure to determine the agreement of EPAD® 2.0 with the conventional intraoperative neurophysiological monitoring.
5. Postoperative focused neurological exam in PACU postoperatively by blinded observer
6. Data analysis/interpretation/presentation/publication

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age>18 years old)
* Scheduled to have either cervical or lumbosacral spine surgery. We include all patients who will undergo either single or multiple instrumented or non-instrumented decompression/fusion with either allograft or autograft bone with a preoperative diagnosis of cervical stenosis, radiculopathy, herniated nucleus pulposus, junctional stenosis, or non-union from prior surgery.

Exclusion Criteria:

* Age <18 years old
* BMI>40
* Unable to perform preoperative neurological examination such as the language barrier
* Fluctuating neurological signs/symptoms (eg. recent CVA, peripheral neuropathy, etc)
* Unable to obtain informed consent
* Contraindication to EP monitoring - skin burns or trauma at EP electrode sites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study Participants: 30 patients who are scheduled to have spine surgery in LHSC.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
The feasibility of using EPAD 2.0 automated device to successfully monitor the patients in spine surgery. | Intraoperative
  The feasibility is determined by the percentage of patients being successfully monitored in spine surgery using the EPAD 2.0 automated device (i.e. [number of patients being successfully monitored/ total number of patients being recruited]*100).

CONTACTS AND LOCATIONS:
Overall Officials: Jason Chui, MBChB, Principal Investigator — University of Western Ontario, Canada

REFERENCES:
- [Background] Ghobrial GM, Williams KA Jr, Arnold P, Fehlings M, Harrop JS. Iatrogenic neurologic deficit after lumbar spine surgery: A review. Clin Neurol Neurosurg. 2015 Dec;139:76-80. doi: 10.1016/j.clineuro.2015.08.022. Epub 2015 Sep 1. PMID 26386902
- [Background] Jimenez JC, Sani S, Braverman B, Deutsch H, Ratliff JK. Palsies of the fifth cervical nerve root after cervical decompression: prevention using continuous intraoperative electromyography monitoring. J Neurosurg Spine. 2005 Aug;3(2):92-7. doi: 10.3171/spi.2005.3.2.0092. PMID 16370297
- [Background] Sasai K, Saito T, Akagi S, Kato I, Ohnari H, Iida H. Preventing C5 palsy after laminoplasty. Spine (Phila Pa 1976). 2003 Sep 1;28(17):1972-7. doi: 10.1097/01.BRS.0000083237.94535.46. PMID 12973145
- [Background] Fan D, Schwartz DM, Vaccaro AR, Hilibrand AS, Albert TJ. Intraoperative neurophysiologic detection of iatrogenic C5 nerve root injury during laminectomy for cervical compression myelopathy. Spine (Phila Pa 1976). 2002 Nov 15;27(22):2499-502. doi: 10.1097/00007632-200211150-00014. PMID 12435981
- [Background] Fehlings MG, Brodke DS, Norvell DC, Dettori JR. The evidence for intraoperative neurophysiological monitoring in spine surgery: does it make a difference? Spine (Phila Pa 1976). 2010 Apr 20;35(9 Suppl):S37-46. doi: 10.1097/BRS.0b013e3181d8338e. PMID 20407350